CLINICAL TRIAL: NCT00816595
Title: Randomized Phase II Trial of Pentostatin, Cyclophosphamide, and Rituximab With or Without Concurrent Avastin® for Previously Untreated B-Chronic Lymphocytic Leukemia (CLL)
Brief Title: Pentostatin, Cyclophosphamide, and Rituximab With or Without Bevacizumab in Treating Patients With B-Cell Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000630491; P30CA015083 (NIH); RC0783 (Registry Identifier: Mayo Clinic Cancer Center); 08-002080 (Other: Mayo Clinic IRB); AVF4491s (Other: Genentech protocol); NCI-2009-01225 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-12-31; First posted 2009-01-01 (Estimated); Results first posted 2014-05-09 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-05

CONDITIONS: Leukemia; Lymphoma
Keywords: B-cell chronic lymphocytic leukemia; stage 0 chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II small lymphocytic lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Bevacizumab; pegfilgrastim; Rituximab; Cyclophosphamide; Pentostatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Pentostatin, Cyclophosphamide, Rituximab, and Avastin (Experimental): Patients receive 15 mg/kg bevacizumab IV over 30-90 minutes on day 1 of courses 1-5 and on days 1, 22, and 43 of course 6; 375 mg/m^2 rituximab IV over 2-4 hours on days 2 and 3 of course 1 and on day 1 of courses 2-6; and 2 mg/m^3 pentostatin IV over 30 minutes and 600 mg/m^2 cyclophosphamide IV over 30 minutes on day 2 of course 1 and on day 1 of courses 2-6. Patients also receive 6 mg pegfilgrastim subcutaneously (SC) on day 3 of course 1 and on day 2 of courses 2-6. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Biological: pegfilgrastim; Biological: rituximab; Drug: cyclophosphamide; Drug: pentostatin
- Arm B: Pentostatin, Cyclophosphamide, and Rituximab (Experimental): Patients receive 100 mg rituximab IV over 2-4 hours on day 1 and 375 mg/m^2 on day 2 of course 1 and 375 mg/m^2 on day 1 of courses 2-6. They receive 2 mg/m^2 pentostatin IV over 30 minutes and 600 mg/m^2 cyclophosphamide IV over 30 minutes on day 1. Patients also receive 6 mg pegfilgrastim SC on day 2. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: pegfilgrastim; Biological: rituximab; Drug: cyclophosphamide; Drug: pentostatin

INTERVENTIONS:
Biological: bevacizumab — Given IV
  Other Names: Avastin
  Arms: Arm A: Pentostatin, Cyclophosphamide, Rituximab, and Avastin
Biological: pegfilgrastim — Given subcutaneously
Biological: rituximab — Given IV
Drug: cyclophosphamide — Given IV
Drug: pentostatin — Given IV

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as pentostatin and cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab and bevacizumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. It is not yet known whether giving pentostatin and cyclophosphamide together with rituximab is more effective with or without bevacizumab in treating patients with B-cell chronic lymphocytic leukemia or small lymphocytic lymphoma.

PURPOSE: This randomized phase II trial is studying the side effects of giving pentostatin and cyclophosphamide together with rituximab with or without bevacizumab and to see how well it works in treating patients with B-cell chronic lymphocytic leukemia or small lymphocytic lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the rate of complete and overall response in patients with B-cell chronic lymphocytic leukemia or small lymphocytic lymphoma treated with pentostatin, cyclophosphamide, and rituximab with or without bevacizumab.
* To assess the proportion of patients who achieve a negative minimal residual disease state after treatment with these regimens.
* To monitor and assess the adverse events of these regimens.

Secondary

* To determine if molecular prognostic parameters (ZAP-70, CD38, cytogenetic abnormalities identified by FISH, and IgVH mutation status) relate to response in these patients.
* To determine the progression-free survival of patients treated with these regimens.
* To complete additional correlative studies to gain insight into disease biology and how it influences drug sensitivity.

OUTLINE: Patients are stratified according to Rai risk group (high [Rai stage III or IV] vs low [Rai stage 0] or intermediate [Rai stage I or II]) and FISH prognosis group (favorable [normal, +12, 13q-, or other] vs unfavorable [17p- or 11q-]). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive bevacizumab IV over 30-90 minutes on day 1 of courses 1-5 and on days 1, 22, and 43 of course 6; rituximab IV over 2-4 hours on days 2 and 3 of course 1 and on day 1 of courses 2-6; and pentostatin IV over 30 minutes and cyclophosphamide IV over 30 minutes on day 2 of course 1 and on day 1 of courses 2-6. Patients also receive pegfilgrastim subcutaneously (SC) on day 3 of course 1 and on day 2 of courses 2-6. Treatment repeats every 21 days* for 6 courses in the absence of disease progression or unacceptable toxicity.

NOTE: *Course 6 is 56 days in duration

* Arm II: Patients receive rituximab IV over 2-4 hours on days 1 and 2 of course 1 and on day 1 of courses 2-6 and pentostatin IV over 30 minutes and cyclophosphamide IV over 30 minutes on day 1. Patients also receive pegfilgrastim SC on day 2. Treatment repeats every 21 days* for 6 courses in the absence of disease progression or unacceptable toxicity.

NOTE: *Course 6 is 56 days in duration

Patients undergo blood sample collection and bone marrow biopsy/aspiration periodically for translational research studies. Samples are analyzed by flow cytometry for assessment of minimal residual disease. Molecular prognostic markers (including CD38, ZAP-70, IgVH gene mutation status, and cytogenetic abnormalities by FISH), Tcl-1 and CD49d protein expression, and immunoglobulin heavy chain D and J family gene usage are also analyzed. Plasma samples are stored for future studies evaluating levels of VEGF, bFGF, and thrombospondin by ELISA.

After completion of study therapy, patients are followed periodically for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Biopsy proven small lymphocytic lymphoma (SLL)
  * Chronic lymphocytic leukemia (CLL)* as evidenced by the following criteria:

    * Peripheral blood lymphocyte count > 5,000/mm³ consisting of small to moderate size lymphocytes
    * Immunophenotyping consistent with CLL, defined by the following:

      * The predominant population of lymphocytes share both B-cell antigens (CD19, CD20, or CD23) as well as CD-5 in the absence of other pan-T-cell markers (CD-3 or CD-2)
      * Dim surface immunoglobulin expression
      * Exclusively kappa and lambda light chains
    * Negative FISH analysis for t(11;14)(IgH/CCND1) on peripheral blood or tissue biopsy samples NOTE: *Splenomegaly, hepatomegaly, or lymphadenopathy are not required for the diagnosis of CLL
* Has ≥ 1 of the following indications** for chemotherapy:

  * Evidence of progressive marrow failure as manifested by the development of or worsening anemia (hemoglobin ≤ 11 g/dL) and/or thrombocytopenia (platelet count ≤ 100,000/mm³)
  * Symptomatic or progressive lymphadenopathy, splenomegaly or hepatomegaly
  * Has ≥ 1 of the following disease-related symptoms:

    * Weight loss > 10% within the past 6 months
    * Extreme fatigue attributed to CLL
    * Fevers > 100.5^oF for 2 weeks without evidence of infection
    * Night sweats without evidence of infection
  * Progressive lymphocytosis (not due to the effects of corticosteroids) with an increase of > 50% over a 2-month period or an anticipated doubling time of < 6 months NOTE: **Marked hypogammaglobulinemia or the development of a monoclonal protein in the absence of any of the above criteria for active disease are not sufficient indications for study treatment

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group performance status 0-3
* Life expectancy ≥ 12 months
* Total bilirubin ≤ 3.0 times upper limit of normal (ULN) (unless due to Gilbert's disease)

  * Direct bilirubin < 1.5 mg/dL (in patients with Gilbert's disease)
* Serum glutamate oxaloacetate transaminase ≤ 3.0 times ULN (unless due to hepatic involvement by CLL)
* Creatinine ≤ 1.5 times ULN
* Urine protein:creatinine ratio < 1.0 OR < 1 g of protein by 24-hour urine collection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 months after completion of study treatment
* Willing to provide mandatory blood and tissue samples
* None of the following cardiovascular conditions:

  * NYHA class III-IV heart disease
  * Myocardial infarction within the past 6 months
  * Unstable angina
  * Stroke, cerebrovascular accident, or transient ischemic attack within the past 6 months
  * Arterial thromboembolic events within the past 12 months
  * Clinically significant peripheral vascular disease
  * Uncontrolled hypertension, defined as systolic BP > 150 mm Hg or diastolic BP > 100 mm Hg

    * Hypertension allowed provided it is controlled with a stable anti-hypertensive regimen
  * History of hypertensive crises or hypertensive encephalopathy
  * Deep venous thromboses or pulmonary embolism within the past 12 months
* No evidence of bleeding diathesis or coagulopathy
* No uncontrolled or active hemolytic anemia requiring immunosuppressive therapy or other pharmacologic treatment
* No active or recent history (within the past 30 days) of hemoptysis (≥ ½ teaspoon of bright red blood per episode)
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No active peptic ulcer disease
* No serious non-healing wound, ulcer, or bone fracture
* No significant traumatic injury within the past 28 days
* No uncontrolled infection
* No active HIV infection
* No other active primary malignancy (except nonmelanoma skin cancer or carcinoma in situ of the cervix) requiring treatment or limiting survival to ≤ 2 years
* No psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude study participation

PRIOR CONCURRENT THERAPY:

* Prior corticosteroids allowed
* More than 4 weeks since prior radiotherapy
* More than 28 days since prior and no concurrent major surgical procedure or open biopsy
* More than 7 days since prior minor surgical procedure, fine needle aspiration, or core biopsy (other than bone marrow biopsy)
* No concurrent therapeutic doses of coumadin-derivative anticoagulants (e.g., warfarin)

  * Doses of ≤ 2 mg daily allowed for prophylaxis of thrombosis
  * Prophylactic doses of low molecular weight heparin allowed
* No other concurrent investigational agents for treatment of CLL or SLL
* No other concurrent specific anticancer treatment except hormonal therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2009-02; Primary Completion 2013-07 (Actual); Study Completion 2016-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tait D. Shanafelt, MD, Study Chair — Mayo Clinic; Jose F. Francisco, M.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Pentostatin, Cyclophosphamide, Rituximab, and Avastin: Patients receive 15 mg/kg bevacizumab IV over 30-90 minutes on day 1 of courses 1-5 and on days 1, 22, and 43 of course 6; 375 mg/m^2 rituximab IV over 2-4 hours on days 2 and 3 of course 1 and on day 1 of courses 2-6; and 2 mg/m^3 pentostatin IV over 30 minutes and 600 mg/m^2 cyclophosphamide IV over 30 minutes on day 2 of course 1 and on day 1 of courses 2-6. Patients also receive 6 mg pegfilgrastim subcutaneously (SC) on day 3 of course 1 and on day 2 of courses 2-6. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  bevacizumab: Given IV pegfilgrastim: Given subcutaneously rituximab: Given IV cyclophosphamide: Given IV pentostatin: Given IV
- Arm B: Pentostatin, Cyclophosphamide, and Rituximab: Patients receive 100 mg rituximab IV over 2-4 hours on day 1 and 375 mg/m^2 on day 2 of course 1 and 375 mg/m^2 on day 1 of courses 2-6. They receive 2 mg/m^2 pentostatin IV over 30 minutes and 600 mg/m^2 cyclophosphamide IV over 30 minutes on day 1. Patients also receive 6 mg pegfilgrastim SC on day 2. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  pegfilgrastim: Given subcutaneously rituximab: Given IV cyclophosphamide: Given IV pentostatin: Given IV
Period: Overall Study
Arm/Group | Arm A: Pentostatin, Cyclophosphamide, Rituximab, and Avastin | Arm B: Pentostatin, Cyclophosphamide, and Rituximab
Started | 35 | 33
Completed | 33 | 33
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Pentostatin, Cyclophosphamide, Rituximab, and Avastin | Arm B: Pentostatin, Cyclophosphamide, and Rituximab | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Continuous [Median (Full Range); unit: years] | 65 [43 to 81] | 63 [50 to 78] | 63.5 [43 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 20 | 24 | 44
Region of Enrollment [Number; unit: participants]
  United States | 33 | 33 | 66

OUTCOME MEASURES:

1. Primary Outcome: Complete and Overall Response Rate
Description: A Complete Response (CR) requires all of the following for 2 months:
  * Absence of lymphadenopathy by physical examination (PE)
  * No hepato- or splenomegaly by PE
  * Neutrophils >1500/ul, Platelets >100,000/ul. Hemoglobin >11.0 gm/dl, Peripheral blood lymphocytes <4000/uL
  Nodular Partial Response (nPR) is defined as a patient qualified for a CR, but regenerative nodules are histologically present on bone marrow samples.
  A Clinical Complete Response (CCR) is defined as a patient qualified for a CR, but bone marrow samples are not available.
  A Partial Response (PR) requires 50% reduction in 2 of the following: peripheral blood lymphocytes, or the sum of the products of the maximal perpendicular diameters, or the size of liver and/or spleen; and a 50% increase in neutrophils, platelets, or hemoglobin.
  Overall response rate is calculated as the number of patients receiving CR, CCR, nPR, or PR as their objective status divided by the total number of evaluable patients.
Time Frame: Evaluated after 6 cycles (up to 196 days)
Population: One patient on Arm A was treated at an incorrect dose level and was not evaluable for this endpoint. On Arm B, one patient did not have correct eligibility reported, one patient did not complete an assessment, and one patient was incorrectly treated. The primary endpoint is based on 32 Arm A and 30 Arm B patients.
Measure: Number; unit: percentage of patients
Arm/Group | Arm A: Pentostatin, Cyclophosphamide, Rituximab, and Avastin | Arm B: Pentostatin, Cyclophosphamide, and Rituximab
Number analyzed (Participants) | 32 | 30
percentage of patients
  Complete Response (CR) Rate | 50.0 | 33.3
  Overall Response Rate | 93.8 | 96.7

2. Secondary Outcome: Overall Survival
Description: The Kaplan-Meier method will be used to estimate overall survival distributions Overall survival is measured as the time from registration to the time of death due to any cause.
Time Frame: Assessed up to 5 years from registration
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Pentostatin, Cyclophosphamide, Rituximab, and Avastin | Arm B: Pentostatin, Cyclophosphamide, and Rituximab
Number analyzed (Participants) | 32 | 30
months | NA [NA to NA] — Insufficient data has been collected to provide an estimate. | NA [54.3 to NA] — Insufficient data has been collected to provide an estimate.

3. Secondary Outcome: Progression-free Survival
Description: The Kaplan-Meier method will be used to estimate progression-free survival distribution. Progression-free survival is defined as the time from registration to the time of progression or death, whichever occurs first.
Time Frame: Assessed up to 5 years from registration
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Pentostatin, Cyclophosphamide, Rituximab, and Avastin | Arm B: Pentostatin, Cyclophosphamide, and Rituximab
Number analyzed (Participants) | 32 | 30
months | NA [26.0 to NA] — Insufficient data has been collected to provide an estimate. | 34.1 [23.0 to 52.1]

ADVERSE EVENTS:
Arm/Group | Arm A: Pentostatin, Cyclophosphamide, Rituximab, and Avastin | Arm B: Pentostatin, Cyclophosphamide, and Rituximab
Serious Adverse Events (participants affected / at risk) | 11/33 | 5/33
Other Adverse Events (participants affected / at risk) | 32/33 | 30/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Pentostatin, Cyclophosphamide, Rituximab, and Avastin (N=33) | Arm B: Pentostatin, Cyclophosphamide, and Rituximab (N=33)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Localized edema (General disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 4 (5) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Bladder hemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis (Renal and urinary disorders) | 2 (2) | 0 (0)
Protein urine positive (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Pentostatin, Cyclophosphamide, Rituximab, and Avastin (N=33) | Arm B: Pentostatin, Cyclophosphamide, and Rituximab (N=33)
Blood disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 13 (52) | 16 (24)
Cardiac disorder (Cardiac disorders) | 2 (4) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (2) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 1 (1) | 1 (1)
Restrictive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (2)
Torsade de pointes (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (7) | 6 (8)
Ascites (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (2)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (16) | 10 (17)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 7 (12) | 6 (11)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 31 (214) | 29 (152)
Fever (General disorders) | 8 (10) | 13 (26)
Hypothermia (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 2 (4)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Immune system disorder (Immune system disorders) | 1 (2) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Gallbladder infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 2 (2)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (5) | 3 (4)
Sepsis (Infections and infestations) | 2 (3) | 3 (4)
Sinusitis (Infections and infestations) | 2 (2) | 1 (2)
Upper aerodigestive tract infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 3 (4) | 6 (9)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 10 (28) | 11 (40)
Neutrophil count decreased (Investigations) | 18 (26) | 17 (36)
Platelet count decreased (Investigations) | 21 (79) | 14 (60)
Weight loss (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 5 (9) | 1 (3)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (1) | 5 (10)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 19 (48) | 11 (23)
Neuralgia (Nervous system disorders) | 1 (1) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2) | 1 (1)
Syncope vasovagal (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (5)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (4) | 1 (4)
Cystitis (Renal and urinary disorders) | 0 (0) | 1 (1)
Hemorrhage urinary tract (Renal and urinary disorders) | 1 (1) | 0 (0)
Protein urine positive (Renal and urinary disorders) | 12 (22) | 3 (3)
Renal failure (Renal and urinary disorders) | 1 (2) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 4 (6) | 2 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (2)
Hot flashes (Vascular disorders) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 17 (52) | 9 (19)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Vascular disorder (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes